CLINICAL TRIAL: NCT01417520
Title: Clinical and Pathophysiological Investigations Into Erdheim-Chester Disease
Brief Title: Clinical and Pathophysiological Investigations Into Erdheim Chester Disease
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110207; 11-HG-0207
Record Dates: First submitted 2011-08-13; First posted 2011-08-16 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07-24

CONDITIONS: Myelofibrosis; Gaucher Disease; Pulmonary Fibrosis; Hermansky-Pudlak Syndrome (HPS); Cancer
Keywords: ECD; Erdheim-Chester Disease
MeSH Terms: conditions — Primary Myelofibrosis; Gaucher Disease; Pulmonary Fibrosis; Hermanski-Pudlak Syndrome; Neoplasms; Erdheim-Chester Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- ECD: ECD patients of any gender and ethnicity age 2-80 years are eligible to enroll in this protocol

SUMMARY:
Background:

- Erdheim Chester Disease (ECD) is a very rare disease in which abnormal white blood cells start growing and affect the bones, kidneys, skin, and brain. ECD can cause severe lung disease, kidney failure, heart disease, and other complications that lead to death. Because ECD is a rare disease, found mostly in men over 40 years of age, there is no standard treatment for it. More information is needed to find out what genes can cause ECD and how best to treat it.

Objectives:

- To collect study samples and medical information on people with Erdheim Chester Disease.

Eligibility:

- Individuals 2 to 80 year of age who have been diagnosed with Erdheim Chester Disease.

Design:

* Participants will be screened with a physical exam and medical history.
* Participants will have a study visit to provide samples for study, including blood, urine, and skin tissue samples. Participants will also have lung, heart, and muscle function tests; imaging studies of the brain, chest, and whole body; a treadmill running stress test; an eye exam; and other tests as needed by the study doctors.
* Participants will be asked to return for a similar set of tests every 2 years, and to remain in contact for possible treatment options.

DETAILED DESCRIPTION:
Rare and potentially lethal, Erdheim-Chester Disease (ECD) is a histiocytic neoplasm about which little is known, and for which there remains a paucity of effective treatments. Histologically, it is categorized as a non-Langerhans cell histiocytosis, and most commonly occurs in men between the ages of 50 and 70, although cases have been reported in women, and rarely, children. Worldwide about 600 cases have been reported, and the disorder remains difficult to diagnose due to its rarity and protean manifestations. The phenotype of ECD ranges from almost asymptomatic patients diagnosed incidentally when imaging studies are done for other reasons, to patients presenting with multiple organ failure who die shortly after diagnosis. These multifarious presentations, and the subsequent response to therapy, have not been well documented and create the need for a prospective study to learn more about this devastating disorder.

Protocol 11-HG-0207, "Clinical and Pathophysiological Investigations into Erdheim-Chester Disease," is a natural history study designed to better understand and describe the natural history, pathophysiology, and response to therapy, of this devastating disorder. We will use a prospective design to enroll and follow qualified men and women, of all ethnic groups, ages 2 to 80 years, who will be screened for candidacy prior to enrollment. If appropriate for the study, patients may opt to be evaluated at the NIH Clinical Center, or may opt to send tissue and records for analysis. The NIH Clinical Center will be the only center for this study, and patients may return for follow-up visits every two to three years, or send copies of test results in lieu of an admission. The enrollment ceiling is 100 patients and we may close the study to new recruitment at that time, but keep the study open to see established patients and to analyze data. Thus, we do not have a definite time-period for the completion of the study.

Through the prospective design, we will collect data from medical histories and physical exams, lab tests, imaging studies, organ-function studies, various measurement tools, and medical consultations. Data will be collated into spreadsheets and divided into functional categories such as organ system complications, to facilitate analysis. We will analyze the data with the assistance of an NIH statistician using parametric and non-parametric methods to assess overall trends in survival, and to look for patterns in organ involvement, patterns in response to various therapeutic regimens, and, lastly, to look for an association between the BRAF V600E mutation and disease severity.

Patient safety and privacy, and respect for the autonomy of the patients, are our top priorities. All patients will be carefully screened prior to participation, and we follow Clinical Center policies regarding informed consent. Data will be stored electronically and in hard copy, in password protected computers and locked cabinets, respectively. Only the PI, the responsible physician, and select AIs, will have access. Patients will be closely monitored during NIH admissions, and the investigators will track all adverse events according to NIH policy. The investigators will keep patients apprised of test results and will reiterate the risks and benefits of procedures during NIH evaluations. Lastly, the investigators will respect patients rights to refuse testing.

We will disseminate the results of our analyses in publications and presentations intended to educate the medical community regarding the diagnosis and management of ECD, and to spur research. We hope our efforts will eventually lead to better outcomes for patients.

ELIGIBILITY:
* INCLUSION CRITERIA:
* ECD patients of any gender and ethnicity age 2-80 years are eligible to enroll in this protocol.
* Patients will be diagnosed as having ECD based upon pathologic evaluations of affected organs.
* Any child older than 2 years with confirmed ECD by pathology will be enrolled in our study since childhood cases are so rare. The child must be clinically stable prior to visiting the NIHCC.
* Patients that agree to be part of this research study are expected to undergo the evaluations and testing of this protocol.

EXCLUSION CRITERIA:

* Patients will be excluded if they have a suspected diagnosis of ECD not confirmed by biopsy or another form of histiocytosis.

  --If the patients cannot travel to the NIH because of their medical condition, they can still participate in our study by submitting tissue and blood for research purposes after consent has been obtained and diagnosis of ECD has been confirmed through tissue-biopsy evaluation. This exception applies to all patients aged 2-80 years.
* Children under age two years are excluded because there is no urgency for a very early diagnosis and care is more readily provided to older children at the Clinical Center.
* Pregnant women will not take part in this study because of the fetal risks, unless they will be participating by only submitting samples of previously collected tissue. We will not encourage pregnant women to undergo affected organ surgery or biopsy to participate in this study, unless clinically indicated and recommended by their private physicians.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2011-08-01; Study Completion 2019-07-24

PRIMARY OUTCOMES:
To comprehensively describe the natural history of ECD, including genetic and epidemiological aspects, its associated complications, and responses to various treatments. | 1 day
  To comprehensively describe the natural history of ECD, including genetic and epidemiological aspects, its associated complications, and responses to various treatments.
To identify molecular markers important for diagnosis and treatment. | 1 day
  To identify molecular markers important for diagnosis and treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J O'Brien, C.R.N.P., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bassou D, El Kharras A, Taoufik AT, En Nouali H, Elbaaj M, Benameur M, Darbi A. Cardiac Erdheim-Chester. Intern Med. 2009;48(1):83-4. doi: 10.2169/internalmedicine.48.1448. Epub 2009 Jan 1. No abstract available. PMID 19122364
- [Background] Aouba A, Georgin-Lavialle S, Pagnoux C, Martin Silva N, Renand A, Galateau-Salle F, Le Toquin S, Bensadoun H, Larousserie F, Silvera S, Provost N, Candon S, Seror R, de Menthon M, Hermine O, Guillevin L, Bienvenu B. Rationale and efficacy of interleukin-1 targeting in Erdheim-Chester disease. Blood. 2010 Nov 18;116(20):4070-6. doi: 10.1182/blood-2010-04-279240. Epub 2010 Aug 19. PMID 20724540
- [Background] Barnes PJ, Foyle A, Hache KA, Langley RG, Burrell S, Juskevicius R. Erdheim-Chester disease of the breast: a case report and review of the literature. Breast J. 2005 Nov-Dec;11(6):462-7. doi: 10.1111/j.1075-122X.2005.00133.x. PMID 16297093